CLINICAL TRIAL: NCT01982669
Title: Effects of Spicy Diet on Salty Taste and Salt Intake
Brief Title: Spicy Diet on Salty Taste and Salt Intake
Status: Completed | Type: Observational
Sponsor: Zhiming Zhu (Other)
Responsible Party: Sponsor-Investigator, Zhiming Zhu, Director of the Dept. of Hypertension & Endocrinology, Third Military Medical University
Organization: Third Military Medical University (Other)
Other Study IDs: SATIETY-1; 2012CB517805 (Other Grant/Funding Number: 973 Program & TMMU Key Clinical Trial Grant)
Record Dates: First submitted 2013-10-27; First posted 2013-11-13 (Estimated); Last update posted 2016-01-11 (Estimated); Status verified 2016-01

CONDITIONS: Salty Taste; Spicy Diet
Keywords: Salty taste; Urinary sodium excretion; Spicy hedonic; Blood pressure

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood, Urine
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Different degree of spicy food intake
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention

SUMMARY:
Excess dietary salt intake is closely associated with the development of hypertension and cardiocerebral vascular diseases. Reduction in high salt intake significantly prevents hypertension and cardiocerebral events. Currently, few promising method is available to reduce salt intake in human. This study focus on examining the salty taste in population-level and exploring whether dietary factors can reduce salt intake through acting on salty taste.

DETAILED DESCRIPTION:
Hypertension and its related complications are common health problems that can lead to multiple organ damage and death. Excessive salt intake plays very important role in the development of hypertension. Reducing salt intake prevents high blood pressure as well as cardiocerebral vascular diseases.

The experimental design is a multi-center, random-order, double-blind observational study to investigate the salty taste and salt intake in population-level.

A total of 606 individuals from four cities in China are recruited in this study. This study aims to explore the salty taste characterization and salt intake in participants who like or dislike spicy diet through questionnaire, spicy preference, salty perception and super-threshold as well as the 24-hour urinary sodium excretion.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years and ≤ 55 years.
* Willing and able to provide written informed consent.
* Willing and able to comply with all study procedures.

Exclusion Criteria:

* Hypogeusia or loss due to neural system disease or oral and digestive disease.
* Capsaicin allergy and poor compliance.
* Recently oral diuretics and participate in other pharmacological experiment in 3 months.
* Acute infection, cancer, serious arrhythmias, drug or alcohol abuse.
* Currently have cold, fever, acidosis, dehydration, diarrhea, vomiting during the study.
* Unwilling or unable to communication due to the dysnoesia and language disorders
* Severe neural or psychiatric diseases that would preclude fully understand and corporation in the study.
* Pregnancy or lactation
* Unwilling to sign the informed consent

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Residents from four cities(Shenyang, Jinan, Chengdu and Chongqing) in China
Sampling Method: Non-Probability Sample
Enrollment: 606 (Actual)
Dates: Start 2013-02; Primary Completion 2013-11 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Effects of spicy diet on salt taste | Day 1
  Daily spicy food intake was evaluated by diet questionnaire and salty taste was tested through salt perception and super-threshold examination on the first day when the participant was investigated.

SECONDARY OUTCOMES:
Effects of spicy diet on salt intake | Day 1
  Daily spicy food intake was evaluated by diet questionnaire on the first day when the participant was investigated and then 24-hour urine was collected during the following day and salt intake was assessed by 24-hour urinary sodium excretion.
Effects of spicy diet on obesity parameters. | Day 1
  Daily spicy food intake was evaluated by diet questionnaire and body mass index and waist circumference were measured on the first day when the participant was investigated.
Effects of spicy diet on blood pressure | Day 1
  Daily spicy food intake was evaluated by diet questionnaire and systolic and diastolic blood pressure were measured on the first day when the participant was investigated.

CONTACTS AND LOCATIONS:
Locations (1):
- Daping Hospital, The Third Military Medical University, Chongqing, Chongqing Municipality, China

REFERENCES:
- [Result] Yang D, Luo Z, Ma S, Wong WT, Ma L, Zhong J, He H, Zhao Z, Cao T, Yan Z, Liu D, Arendshorst WJ, Huang Y, Tepel M, Zhu Z. Activation of TRPV1 by dietary capsaicin improves endothelium-dependent vasorelaxation and prevents hypertension. Cell Metab. 2010 Aug 4;12(2):130-41. doi: 10.1016/j.cmet.2010.05.015. PMID 20674858
- [Result] Zhang LL, Yan Liu D, Ma LQ, Luo ZD, Cao TB, Zhong J, Yan ZC, Wang LJ, Zhao ZG, Zhu SJ, Schrader M, Thilo F, Zhu ZM, Tepel M. Activation of transient receptor potential vanilloid type-1 channel prevents adipogenesis and obesity. Circ Res. 2007 Apr 13;100(7):1063-70. doi: 10.1161/01.RES.0000262653.84850.8b. Epub 2007 Mar 8. PMID 17347480
- [Result] Hao X, Chen J, Luo Z, He H, Yu H, Ma L, Ma S, Zhu T, Liu D, Zhu Z. TRPV1 activation prevents high-salt diet-induced nocturnal hypertension in mice. Pflugers Arch. 2011 Mar;461(3):345-53. doi: 10.1007/s00424-011-0921-x. Epub 2011 Jan 19. PMID 21246380